CLINICAL TRIAL: NCT06968572
Title: A Phase I, Open-label, Dose-escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic of HSK41959 in Patients With MTAP Deletion Locally Advanced or Metastatic Solid Tumors
Brief Title: Phase I Study of HSK41959 in Solid Tumors With MTAP Deletion
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK41959-101
Record Dates: First submitted 2025-04-09; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase Ia (Part A): HSK41959 as monotherapy (Experimental): Phase 1a (Part A): dose escalation of HSK41959 as monotherapy at various dose levels
  Interventions: Drug: HSK41959
- Phase Ia (Part B): HSK41959 as monotherapy (Experimental): Phase 1a (Part B): dose extention of HSK41959 as monotherapy at certain dose levels
  Interventions: Drug: HSK41959
- Phase Ib: HSK41959 as monotherapy (Experimental): Phase 1b: dose expansion for HSK41959 as monotherapy at a dose determined during Phase 1a (Part B) in patients with MTAP Deletion locally advanced or metastatic solid tumors
  Interventions: Drug: HSK41959

INTERVENTIONS:
Drug: HSK41959 — Oral administration, QD

SUMMARY:
This is a phase I, open-label, dose-escalation and expansion study to evaluate the safety, tolerability, PK and PD of HSK41959 when given orally in patients with MTAP Deletion locally advanced or metastatic Solid Tumors.

DETAILED DESCRIPTION:
The study will contain two phases: Phase Ia is dose escalation phase and Phase Ib is dose expansion phase.

Phase Ia will contain two part: Dose Escalation Part (Part A) and Extension Part (Part B). Part A based on the "3+3" design for dose escalation and safety evaluation requirements. Patient cohorts at selected doses may be extended to further investigate the tolerability, PK and PD of HSK41959. The number of patients to be enrolled will be up to 10 subjects in each Part B cohort. Approximately 30-50 subjects will be enrolled in Phase Ia.

Phase Ib no less than 10-50 subjects will be enrolled in each expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years，Male and female patients, at time of signing informed consent form (ICF).
2. ECOG performance status 0-1.
3. Life expectancy ≥ 3 months.
4. Patients with locally advanced or metastatic solid tumors confirmed by histology or cytology, who have failed standard treatment (disease progression after treatment or intolerable treatment).
5. Homozygous deletion of the MTAP gene detected in tumor tissue confirmed prior to the administration of HSK41959.
6. Measurable disease by RECIST 1.1 criteria.
7. Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

1. Prior treatment with a PRMT5 or MAT2A inhibitor therapy.
2. The presence of unstable, clinically symptomatic central nervous system metastases or leptomeningeal metastases.
3. Malignant tumor within 2 years, with the exception of cutaneous squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma, or other tumors with low malignancy.
4. Uncontrollable pleural effusion, ascites, or pericardial effusion per protocol.

   Treatment with any of the following:
5. Prior treatment with anti-tumor drug within 4 weeks or approximately 5 × t1/2 prior to the first dose of HSK41959, whichever is shorter; Prior treatment with nitrosourea or mitomycin C within 6 weeks prior to the first dose of HSK41959; Prior treatment with palliative radiotherapy or anti-tumor herbs within 2 weeks prior to the first dose of HSK41959; Prior treatment with radiotherapy, electric field therapy, or other anti-tumor therapies within 4 weeks prior to the first dose of HSK41959.
6. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment, with the exception of alopecia, dermal toxicity, and other toxicity considering no safety risks by investigator.
7. Any disease which would preclude drug absorption, metabolism or pharmacokinetics, e.g. active peptic ulcer or chronic gastroesophageal reflux disease.
8. Patients who have clinically significant or uncontrolled cardiac disease, include: QTc interval ≥ 450(male)/470(female) msec; any clinically significant arrhythmia; left ventricular ejection fraction < 50%; myocardial infarction, unstable angina, or class III/IV cardiac failure by the NYHA that occurred within 6 months prior to the first dose of HSK41959.
9. Any thromboembolic events within 6 months prior to the first dose of HSK41959; any familial or acquired thrombophilia.
10. Uncontrolled hypertension (systolic pressure≥160mmHg, or diastolic pressure≥100mmHg), diabetes (fasting blood-glucose≥10mmol/L), seizures, chronic obstructive pulmonary disease (COPD), interstitial pneumonia, pulmonary interstitial fibrosis, Parkinson's disease, active bleeding, or systemic active infection.
11. Any unstable systemic disease, e.g. severe metabolic disease: liver cirrhosis, renal failure, or uremia.
12. Patient with cognitive dysfunction, or history of mental illness, other uncontrolled comorbidities, alcohol dependence, hormone dependence or drug abuse.
13. Other protocol-defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2028-05-08 (Estimated)

PRIMARY OUTCOMES:
DLTs | 24 days
  Incidence of dose-limiting toxicities (DLTs) at Cycle 0 and Cycle1
MTD | 24 days
  MTD determination: dose limiting toxicity (DLT) rate
AEs | Up to approximately 3 years
  Rate and severity of adverse events of HSK41959 as monotherapy
RP2D | Up to approximately 1 year
  RP2D determination: DLT, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary safety and anticancer activity data

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 3 years
  ORR, defined as the proportion of patients who experience a best response of confirmed CR or PR according to RECIST 1.1
Disease control rate (DCR) | Up to approximately 3 years
  DCR, defined as the proportion of patients who experience a best response of CR, PR, or stable disease (SD) according to RECIST 1.1
Duration of response (DOR) | Up to approximately 3 years
  DOR, defined as the time from first documented response of complete response (CR) or partial response (PR) to the date of first documented progressive disease or death due to any cause, whichever occurs first
Progression free survival (PFS) | Up to approximately 3 years
  PFS, defined as the time frocease or death due to any cause, whichever occurs first
Overall survival (OS) | Up to approximately 3 years
  OS, defined as the time from the first dose of HSK41959 until the date of death due to any cause
Area under the curve (AUC) of HSK41959 | Up to approximately 6 months
maximum plasma concentration (Cmax) of HSK41959 | Up to approximately 6 months
half-life (t1/2) of HSK41959 | Up to approximately 6 months
Tmax(Time to maximum plasma concentration) of HSK41959 | Up to approximately 6 months

OTHER OUTCOMES:
Changes in SDMA concentration | Up to approximately 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Shanghai East Hospital, Shanghai, Shanghai Municipality